CLINICAL TRIAL: NCT04114955
Title: Reducing Intersectional Stigma Among High-Risk Women in Brazil to Promote Uptake of HIV Testing and PrEP
Acronym: PRISM Brazil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Santa Casa Medical School (Other); National Institute of Mental Health (NIMH) (NIH); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: R01MH121308 (NIH); R01MH121308 (NIH)
Record Dates: First submitted 2019-09-24; First posted 2019-10-03 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: HIV Prevention
Keywords: transgender women; HIV prevention; HIV testing; pre-exposure prophylaxis; Brazil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Intervention condition comprised of two components designed to address intersectional stigma: 1) a group-level, peer-led intervention and 2) an individual-level peer navigation program to increase uptake of HIV testing and PrEP.
  Interventions: Behavioral: Manas por Manas
- Wait-list control (Other): Control participants will receive the intervention after a one-year waiting period.
  Interventions: Behavioral: Manas por Manas

INTERVENTIONS:
Behavioral: Manas por Manas — Manas for Manas works at both the group- and individual-levels to increase self-care and reduce the negative health impacts of stigma, including: 1) a group-level, peer-led intervention, which first demonstrated efficacy with trans women in the US as 'Sheroes' and has been successfully adapted for Brazil, and 2) an individual-level peer navigation program.

SUMMARY:
This is a randomized controlled trial of a multi-level intervention to prevent HIV acquisition among transgender women (N=400) in São Paulo, Brazil. The intervention will be evaluated using a randomized wait-list controlled trial to compare uptake of HIV testing (self-testing and clinic-based) (Aim 1), PrEP initiation and persistence (Aim 2), and other prevention services (e.g. harm reduction) among trans women in the intervention arm compared to those in the control arm with data collection scheduled every three-months. Investigators will assess changes in intersectional stigma (Aim 3), including reductions in internalized stigma and increased resilience to anticipated and enacted stigma, among those assigned to intervention compared to those assigned to the control arm, and assess how changes in stigma result in prevention uptake.

DETAILED DESCRIPTION:
Globally, transgender ('trans') women experience extreme social and economic marginalization due to intersectional stigma, defined as the confluence of stigma that results from the intersection of social identities and positions among those who are multiply oppressed. Among trans women, gender-based stigma intersects with social positions such as engagement in sex work and substance use, generating a social context of vulnerability and increased risk of HIV acquisition. In Brazil, trans women are the 'most-at-risk' group for HIV, with 55 times higher estimated odds of HIV infection than the general population; further, uptake of HIV testing and pre-exposure prophylaxis (PrEP) among trans women is significantly lower than other at-risk groups, despite availability in the public sector and documented interest in the community. Through extensive formative work, the investigators have developed a suite of evidence-informed interventions and HIV prevention strategies, all of which have demonstrated feasibility and acceptability by trans women in Brazil, to address intersectional stigma and increase engagement of trans women in the HIV prevention continuum. We propose to test a multi-level intervention, 'Guerreiras' ('warrior women', as named by trans women participants in Brazil), comprised of two intervention components designed to address intersectional stigma: 1) a group-level, peer-led intervention and 2) an individual-level peer navigation program to increase uptake of HIV testing and PrEP. Guerreiras is informed by a trans-specific conceptual model, gender affirmation theory, that describes intersectional stigma faced by trans women and frames investigations of how intersectional stigma results in health disparities, providing a framework for the development and testing of interventions to address intersectional stigma among trans women. The study team will recruit trans women (N=400) from clinical sites, outreach events, and an ongoing observational cohort in São Paulo, Brazil. Guerreiras will be evaluated using a randomized wait-list controlled trial to compare uptake of HIV testing (self-testing and clinic-based) (Aim 1), PrEP initiation and persistence (Aim 2), and other prevention services (e.g. harm reduction) among trans women in the intervention arm compared to those in the control arm with data collection scheduled every three-months. Investigators will assess changes in intersectional stigma (Aim 3), including reductions in internalized stigma and increased resilience to anticipated and enacted stigma, among those assigned to intervention compared to those assigned to the control arm, and assess how changes in stigma result in prevention uptake. Outcomes will be monitored through the national medications dispensing system (PrEP initiation and persistence), through clinical records and self-report (HIV testing), and through comprehensive surveys (intersectional stigma). The proposed research leverages a productive multi-disciplinary HIV research partnership with extensive experience working with trans women in Brazil, multi-level intervention components, and a context where PrEP and HIV Self Tests are available publicly, providing an opportunity to evaluate and scale-up an HIV prevention initiative in a key health disparity population, while contributing to nascent research in intersectional stigma.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* assigned 'male' at birth but currently identify as female, transgender, transsexual, or travesti (a common identity term among trans women in Brazil);
* not be known to be HIV positive;
* be a resident of the São Paulo area; and
* consent to study procedures, including consent to review their clinical records.

Exclusion Criteria:

* currently psychotic, suicidal, or manic;
* known to be HIV-positive at enrollment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Assigned 'male' at birth but currently identify as female, transgender, transsexual, or travesti (a common term for trans women in Brazil)
Enrollment: 392 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Changes in HIV testing | Every 3 months through study completion, up to 12 months
  Self- and clinic-based HIV testing
Changes in PrEP uptake | Every 3 months through study completion, up to 12 months
  Initiation of pre-exposure prophylaxis, measured as first filled PrEP prescription
Changes in PrEP persistence | Every 3 months through study completion, up to 12 months
  Persistence of pre-exposure prophylaxis, measured as sufficient pill dispensation for complete 3-month coverage with no more than 10 days uncovered in the period

SECONDARY OUTCOMES:
Changes in PrEP adherence | Every 3 months through study completion, up to 12 months
  Drug levels; Dried blood spots
Changes in condom use | Every 3 months through study completion, up to 12 months
  Self-reported consistent condom use with regular and occasional partners and clients
Changes in utilization of sexual health services | Every 3 months through study completion, up to 12 months
  Clinical data extraction

CONTACTS AND LOCATIONS:
Overall Officials: Jae Sevelius, PhD, Principal Investigator — University of California, San Francisco; Columbia University; Sheri Lippman, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- Brazil (2):
  - CRT - Centro de Referência e Treinamento DST/AIDS, São Paulo
  - SAE - Serviço de Assistência Especializada Campos Elíseos, São Paulo

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/55/NCT04114955/ICF_000.pdf